CLINICAL TRIAL: NCT06625398
Title: REVEAL-2 - A Phase 3, Randomized, Double-masked, Placebo-controlled, Efficacy, Safety, and Tolerability Study of VRDN-003 in Participants With Chronic Thyroid Eye Disease (TED)
Brief Title: An Efficacy, Safety, and Tolerability Study of VRDN-003 in Participants With Chronic Thyroid Eye Disease (TED)
Acronym: REVEAL-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VRDN-003-302
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Eye Disease
Keywords: TED; Thyroid Eye Disease; Graves; Thyroid-Associated Ophthalmopathy; Dysthyroid Ophthalmopathy; Graves Eye Disease; Graves Orbitopathy; Myopathic Ophthalmopathy; Edematous Ophthalmopathy; Infiltrative Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the three study arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to one of the three study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- VRDN-003 every 4 weeks (Experimental): 6 subcutaneous administrations of VRDN-003
  Interventions: Drug: VRDN-003
- VRDN-003 every 8 weeks (Experimental): 3 subcutaneous administrations of VRDN-003 and 3 subcutaneous administrations of placebo
  Interventions: Drug: VRDN-003; Drug: Placebo
- Placebo every 4 weeks (Placebo Comparator): 6 subcutaneous administrations of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VRDN-003 — VRDN-003 is an investigational, subcutaneously administered, humanized monoclonal antibody directed against the Insulin-like Growth Factor-1 receptor (IGF-1R).
  Arms: VRDN-003 every 4 weeks; VRDN-003 every 8 weeks
Drug: Placebo — All participants will receive the same number of injections to maintain masking. Masking will be maintained by the use of placebo injections that appear identical to VRDN-003 injections.
  Arms: Placebo every 4 weeks; VRDN-003 every 8 weeks

SUMMARY:
This is a clinical trial assessing the efficacy, safety, and tolerability of an investigational drug, VRDN-003, in participants with chronic Thyroid Eye Disease (TED).

DETAILED DESCRIPTION:
This is a randomized (meaning participants will be assigned to study arms by chance), double-masked (meaning study doctor and participant will not know which study arm participant is assigned to), placebo-controlled study that will include participants with chronic TED. The key objectives of this study are to determine if VRDN-003 is efficacious, safe and tolerable when administered as subcutaneous/SC injections every 4 weeks or every 8 weeks compared to placebo in participants with chronic TED.

Participants who do not have a meaningful response at Week 24 (irrespective of the initial treatment arm) may be eligible to receive additional subcutaneous injections of VRDN-003.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have moderate to severe chronic TED, with any CAS (0-7) on the 7-item scale, and with documented evidence of ocular symptoms or signs that began greater than 15 months prior to screening
* Must agree to use highly effective contraception as specified in the protocol
* Female TED participants must have a negative serum pregnancy test at screening

Key Exclusion Criteria:

* Must not have received prior treatment with another anti-IGF-1R therapy
* Must not have received systemic corticosteroids or steroid eye drops for any condition, including TED, or selenium within 2 weeks prior to first dose.
* Must not have received other immunosuppressive drugs for any condition, including TED, or any other therapy for TED within 12 weeks prior to first dose
* Must not have received an investigational agent for any condition, including TED, within 8 weeks or longer duration (depending on the type of investigational agent) prior to first dose
* Must not have received radioactive iodine (RAI) treatment within 8 weeks prior to first dose
* Must not have had previous orbital irradiation or decompression surgery for TED to the study eye's orbit
* Must not have a pre-existing ophthalmic condition in the study eye which in the study doctor's opinion, would interfere with interpretation of study results
* Must not have abnormal hearing test before first dose. Must also not have a history of ear conditions considered significant by study doctor
* Must not have a history of inflammatory bowel disease
* Female TED participants must not be pregnant or breastfeeding

NOTE: There are additional eligibility criteria for participants who do not have a meaningful response at Week 24 (irrespective of initial treatment arm) who may receive additional injections of VRDN-003. These are described in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Title: Proptosis Responder Rate in the study eye | At Week 24
  Description: Proportion of participants with a ≥2 mm reduction from baseline in proptosis in the study eye [without a corresponding increase of ≥2 mm in the fellow eye]

SECONDARY OUTCOMES:
Change from baseline in proptosis in the study eye | At Week 24
  Change from baseline in proptosis in the study eye
Overall Responder Rate in the study eye | At Week 24
  Proportion of participants with a ≥2 mm reduction from baseline in proptosis in the study eye [without a corresponding increase of ≥2 mm in the fellow eye] AND no worsening in CAS from baseline in the study eye [without a corresponding increase of ≥2 points in the fellow eye]
Diplopia Responder Rate for participants with baseline Diplopia Score greater than 0 | At Week 24
  Proportion of participants with a reduction in Diplopia Score of ≥1 from baseline (for participants with baseline Diplopia Score greater than 0)
Diplopia Resolution Rate for participants with baseline Diplopia Score greater than 0 | At Week 24
  Proportion of participants with a reduction in Diplopia Score to 0 from baseline (for participants with baseline Diplopia Score greater than 0)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (37):
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Alliance Research Institute - Canoga Park, Canoga Park, California
  - Marvel Clinical Research, Huntington Beach, California
  - United Medical Research Institute, Inglewood, California
  - Advancing Research International, LLC, Los Angeles, California
  - Roski Eye Institute, Keck School of Medicine, USC, Los Angeles, California
  - Alliance Research Institute - Lynwood, Lynwood, California
  - A.P.J. Office, Newport Beach, California
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Pasadena Clinical Trials, Pasadena, California
  - Senta Clinic, San Diego, California
  - Ilumina Medical Research, Kissimmee, Florida
  - Med-Care Research, Miami, Florida
  - Hype Clinical Research LLC, Miami, Florida
  - Anmed Health Services LLC, Miami, Florida
  - Southern Clinical Research LLc, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Vision Medical Research, Orland Park, Illinois
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Opthalmic Consultants of Boston, East Weymouth, Massachusetts
  - Fraser Eye Care Center, Fraser, Michigan
  - Kahana Oculoplastic & Orbital Surgery, Livonia, Michigan
  - University Health, Kansas City, Missouri
  - S.L. Office, Las Vegas, Nevada
  - Vector Clinical Trials, Sparks, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Asheville Clinical Research, Asheville, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Scheie Eye Institute Penn Presbyterian, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Horizon Clinical Research Group, Cypress, Texas
  - Baylor College of Medicine/Alkek Eye Center, Houston, Texas
  - Gulf Coast Clinical Trials, Houston, Texas
  - Neuro-Eye Clinical Trials, Houston, Texas
  - University of Washington, Eye institute, Seattle, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia